CLINICAL TRIAL: NCT07360860
Title: Comparison Between Efficacy and Safety of PRP With Microneedling and Microneedling Alone in Treatment of Macular Amyloidosis; a Split Face Blinded Non Randomized Control Trial With Dermoscopic and Histopathologic Evaluation
Brief Title: Microneedling Alone vs Microneedling With PRP in the Treatment of Macular Amyloidosis; a Split Face Comparative Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Elbendary, Lecturer in Cairo University, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS-59-2025
Record Dates: First submitted 2025-12-27; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Macular Amyloidosis
Keywords: Macular amyloidosis; Microneedling; PRP
MeSH Terms: interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Face split
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- microneedling (Active Comparator): microneedling will be done on the first arm
  Interventions: Device: microneedling
- macular amyloidosis treated with microneedling and PRP (Active Comparator)
  Interventions: Device: microneedling with PRP

INTERVENTIONS:
Device: microneedling — microneedling will be done for the one arm of macular amyloidosis
  Arms: microneedling
Device: microneedling with PRP — microneedling with PRP will be done on macular amyloidosis
  Arms: macular amyloidosis treated with microneedling and PRP

SUMMARY:
This study is going to asses and compare the efficacy of treatment of macular amyloidosis using microneedling vs PRP with microneedling. Pruritus and pigmentation will be assessed.

ELIGIBILITY:
Inclusion Criteria: • Both genders were included.

* Patients above 18 years old.
* Patients diagnosed by macular amyloidosis, proved by dermoscopy and histopathology.

Exclusion Criteria: • Prior use of topical therapies in the previous 4 weeks.

* Prior use of any procedures such as chemical peel or laser treatment in the previous 1 month.
* Prior use of any systemic treatment for macular amyloidosis in the past 12 weeks.
* Patients with other skin conditions (e.g., psoriasis, eczema).
* Immunocompromised patients (HIV, chemotherapy).
* Patients with history of any type of autoimmune disorders, coagulopathies, and keloid tendency.
* Known or suspected allergy to ingredients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement of macular amyloidosis using microneedling or PRP with microneedling | 3 months
  1. The clinical assessment will be performed based on the photographs taken at baseline, after 1month, and 3 months of the last session.
  2. Results will be measured by the Quartile grading scale:
  1< 25% improvement 2=25-<50% improvement 3=50-<75% improvement 4> 75% improvement 3. Degree of improvement in dermoscopic features will be measured by scoring system as follows : 0-25% = 0 (no improvement) 26-50% = 1(mild improvement) 51-75% = 2 (moderate improvement) 76- 100% = 3 (marked improvement) 4. Patients' satisfaction: Visual Analog Score for pain 5.measuring the Treatment Satisfaction Questionnaire for Medication (TSQM) for effectiveness.
  6. TPhysician global satisfaction will be assessed. 0-3 (unsatisfied) 4-6 (satisfied) 7-10 (highly satisfied)

IPD SHARING:
Plan to Share IPD: No